CLINICAL TRIAL: NCT06871124
Title: Early Neuromodulation for Cognitive Recovery and Rehabilitation in Traumatic Brain Injury
Brief Title: Early Neuromodulation in Traumatic Brain Injury
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Cincinnati (Other)
Responsible Party: Principal Investigator, Ishita Basu, Assistant Professor, University of Cincinnati
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TP230311; TP230311 (Other Grant/Funding Number: DOD-CDMRP)
Record Dates: First submitted 2025-02-27; First posted 2025-03-11 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Traumatic Brain Injury (TBI) Patients
Keywords: transcranial electrical stimulation; cognitive control; working memory; EEG
MeSH Terms: conditions — Brain Injuries, Traumatic | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Early intervention (Experimental): Patients assigned to this arm will receive anodal transcranial electrical stimulation (A-tES) within a 1-2 weeks of their injury and another session of tES at a 3 month follow up visit.
  Interventions: Device: transcranial electrical stimulation
- Sham (Sham Comparator): Patients assigned to this arm will receive sham transcranial electrical stimulation (tES) within a 1-2 weeks of their injury and another session of tES at a 3 month follow up visit.
  Interventions: Device: Sham Comparator

INTERVENTIONS:
Device: transcranial electrical stimulation — Anodal transcranial electrical stimulation (A-tES) is a widely used and well tolerated non-invasive electrical stimulation paradigm that promotes adaptive neuroplasticity and may prevent or reduce pathological sequela following brain injury. It has been used in a wide variety of neurologic and psychiatric disorders for cognitive and motor rehabilitation.
  Arms: Early intervention
Device: Sham Comparator — Sham comparator consist of A-tES in the beginning and end of stimulation block but no stimulation during the actual stimulation period.
  Arms: Sham

SUMMARY:
The two goals of the proposed study are: (1) To determine how brain activity changes with cognitive recovery over time from acute to chronic phases of traumatic brain injury (TBI). (2) To determine how the time of anodal transcranial electrical stimulation (A-tES) administration affects cognitive performance and brain activity in TBI.

To achieve these study goals, the investigators will conduct a pilot clinical trial over three years in which the investigators aim to recruit 60 patients with moderate to severe TBI at the University of Cincinnati Medical Center (UCMC). During the acute phase of TBI, all participants will complete clinical questionnaires and perform 2 cognitive computer tasks while their brain activity is recorded. Half of the participants will be randomly selected to receive A-tES for 15 minutes while performing cognitive tasks and the other half will receive sham stimulation. All participants will be followed for 6 months. During their 3-month follow-up, the investigators will perform another session where all participants complete the questionnaires and receive A-tES while performing cognitive tasks during brain recording. In their last visit at 6 months post-injury, all participants will complete the questionnaires and cognitive tasks with brain recording but no stimulation treatment. From the collected data, the investigators will determine if time from brain injury correlates with brain activity during performance of cognitive tasks. The investigators will also assess the efficacy of early A-tES treatment for improving cognitive task performance and clinical test ratings at 6 months post-injury in comparison to A-tES delivered during the 3-month follow-up visit.

DETAILED DESCRIPTION:
Background: Traumatic Brain Injury (TBI) is a medical and surgical epidemic affecting at least 1.7 million individuals yearly in the United States. Functional outcomes after TBI can show improvement or deterioration up to two decades after injury, and rates of all-cause mortality remain elevated for many years. Cognitive impairments are among the most disabling of post-TBI symptoms and typically contribute more to persisting disability than physical impairment. Following TBI, deficits are consistently demonstrated in the domains of attention, working memory and executive functioning. To date, there are some potential interventions for motor/functional recovery but there is no treatment for cognitive dysfunction which is more disabling. Although brain stimulation techniques appear promising as treatments to improve neuropsychiatric conditions and functional deficits, most noninvasive brain stimu¬lation interventions have been nontargeted and focused on the chronic phase of recovery after TBI. In the acute stages, there is limited available evidence of the efficacy and safety of brain stimulation to improve outcomes. The stimulation during chronic phase is applied either in isolation or before cognitive training. TBI thus underscores a major unaddressed challenge: the lack of time sensitive cognitive rehabilitation therapy post injury. Thus, there is an urgent need to develop rehabilitation paradigms in the early phases of injury for cognitive recovery and prevention of long-term cognitive impairments.

Hypothesis/Objective(s): This study is based on the hypothesis that early intervention with anodal transcranial electrical stimulation (A-tES) during the acute and sub-acute phases of TBI will enhance cognitive recovery over a similar intervention used only in the sub-acute phase. The objective of this study is to determine neural biomarkers of cognitive functional recovery in TBI and to investigate the neuromodulatory effects of early A-tES on cognitive functions in the sub-acute/chronic phases of TBI.

Specific Aims: (1) To determine neural correlates of cognitive recovery from injury over the acute to sub-acute/chronic phase in TBI, (2) To determine effects of time from injury when A-tES was administered on cognitive performance and associated EEG rhythms in TBI.

Study Design: The investigators will conduct a pilot clinical trial over a 3-year period in which we aim to recruit 60 patients with moderate to severe isolated TBI at the University of Cincinnati Medical Center (UCMC). All recruited participants will be administered a Brief test of adult cognition (BTACT) at bedside during the acute phase. They will perform 2 cognitive tasks on a laptop computer while their EEGs are being recorded. 50% of recruited patients selected randomly during the acute phase will receive active A-tES to their left dorsolateral prefrontal cortex (dlPFC) for 15 minutes each during the performance of cognitive tasks while the rest will receive sham stimulation. All participants will be followed for 6 months. When they return for their typical 3-month follow-up, we will perform another session with BTACT, EEG and cognitive tasks. During this visit all participants will receive active A-tES to their left dlPFC while performing cognitive tasks. In their last visit at 6 months post injury, all participants will be administered BTACT and cognitive tasks with EEG recordings but no intervention. They will also complete a quality of life (QOL) questionnaire designed through involvement of CBPR during their follow-up visits. For Aim 1, the investigators will determine if there are significant temporal correlations between neural oscillations recorded via EEG during the performance of cognitive tasks and injury phase. For Aim 2, the investigators will use a double-blind, randomized, sham-controlled, parallel study design to assess effects of early A-tES on improving performance on computer tasks, clinical test ratings and QOL measures during the 6-month post injury follow-up compared to A-tES delivered during the 3-month follow up visit.

ELIGIBILITY:
Inclusion Criteria:

1. Moderate to severe TBI: Glasgow Coma Scale (GSC) in the 3-12 range and greater than 30 min of loss of consciousness and/or a post-traumatic amnesia that lasts more than 24 hours and/or an alteration of mental state over 24 hours,
2. age 18-80 years,
3. Isolated TBI,
4. Intelligible speech and Galveston Orientation and Amnesia Test (GOAT) score >70 at time of enrollment.

Exclusion Criteria:

1. Persistent bilateral non-reactive pupils or other evidence of non-survivable injury,
2. Decompressive craniectomy to treat refractory ICP subsequent to diffuse injury, (3) Co-enrollment in another therapeutic TBI trial,

(4) Pregnancy, (5) Patients with polytrauma (6) Patients with clinical seizures or status epilepticus.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-06-16 (Estimated); Primary Completion 2027-09-30 (Estimated); Study Completion 2027-11-30 (Estimated)

PRIMARY OUTCOMES:
Cognitive Task Behavior | from enrollment to 6 months after brain injury
  Response time and accuracy on multi source interference task and 1-back working memory task.
Task evoked EEG oscillatory power | from enrollment to end of 6 month visit
  Task evoked theta and alpha band power

SECONDARY OUTCOMES:
Brief Test of Adult Cognition by Telephone (BTACT) | from enrollment to 6 months after brain injury
  The Brief Test of Adult Cognition by Telephone (BTACT) assesses multiple dimensions central for effective functioning across adulthood: episodic memory, working memory, reasoning, verbal fluency, and executive function. The BTACT is the first instrument which includes measures of processing speed, reaction time, and task switching/inhibitory control for use over the telephone.
Quality of Life (QOL) | from enrollment to 6 months after brain injury
  We will formulate a QOL by partnering with a community advisory board comprising of TBI survivors and their caregiver/family members.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Cincinnati, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: Undecided